CLINICAL TRIAL: NCT06666855
Title: A Phase III Study Including a Single-Arm, Open-Label, Multi-Dose PK Study Cohort and a Randomized, Evaluator-Masked, Active Drug Controlled, Parallel Group, Multicenter, Bridging Study Cohort With a Long-term Follow-up Phase Assessing the Efficacy and Safety of DE-117B Eye Drops in Subjects With Primary Open Angle Glaucoma or Ocular Hypertension in China
Brief Title: A Phase III Study in Subjects With Primary Open Angle Glaucoma or Ocular Hypertension in China
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0117B02CN
Record Dates: First submitted 2024-10-29; First posted 2024-10-31 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DE-117B Eye Drops (Experimental): 0.002% DE-117B Eye Drops - One drop daily, 9:00 PM±1 hours instilled in both eyes for 4 weeks, followed by 0.002% DE-117B Eye Drops - One drop daily, 9:00 PM±1 hours instilled in both eyes for an extension follow-up phase of 12 months.
  Interventions: Drug: DE-117B Eye Drops
- Latanoprost Eye Drops (Active Comparator): 0.005% Latanoprost Eye Drops - One drop daily, 9:00 PM±1 hours instilled in both eyes for 4 weeks, followed by 0.002% DE-117B Eye Drops - One drop daily, 9:00 PM±1 hours instilled in both eyes for an extension follow-up phase of 12 months.
  Interventions: Drug: Latanoprost

INTERVENTIONS:
Drug: DE-117B Eye Drops — Investigational Product: 0.002% DE-117B Eye Drops
  Arms: DE-117B Eye Drops
Drug: Latanoprost — Active Control: 0.005% Latanoprost Eye Drops
  Arms: Latanoprost Eye Drops

SUMMARY:
This is a Phase III Study that includes a single arm, open-label, multi-dose PK study cohort and a randomized, evaluator-masked, active drug-control multicenter study.

Subjects diagnosed with POAG (Primary Open Angle Glaucoma) or OHT (Ocular Hypertension) who meet eligibility criteria will washout of their current IOP lowering medication(s), if any.

The study will investigate plasma pharmacokinetics of multi-dose 0.002% DE-117B eye drops (1 drop at a time administered once daily for 7 days) in Chinese subjects with primary open angle glaucoma or ocular hypertension.

It will investigate the safety of multi-dose 0.002% DE-117B eye drops (1 drop at a time administered once daily for 7 days) in Chinese subjects with primary open angle glaucoma or ocular hypertension.

There will be a bridging cohort and extension follow-up phase

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with primary open angle glaucoma or ocular hypertension in both eyes.
* Corrected visual acuity ≥0.2 in both eyes.
* Anterior chamber angle grade ≥2 (Shaffer scale) in both eyes.
* Central corneal thickness ≥480 μm to ≤600 μm in both eyes.
* At completion of the washout phase, IOP ≥22 mmHg in at least one eye and ≤34 mmHg in both eyes at all measurement time points.

Exclusion Criteria:

* Consider visual field disorder at risk for progression during the study based on the current clinical examination result.
* Severe visual field disorder (e.g., mean deviation lower than -12 dB, as assessed by Humphrey field analyzer).
* Any corneal abnormality or other condition potentially interfering with reliable applanation tonometry.
* History of iritis or uveitis.
* Presence of any active external ocular disease, inflammation, or infection of the eye or eyelids.
* History of macular oedema, retinal detachment, or diabetic retinopathy, or current retinal disease at risk for progression during the study.
* History of refractive keratotomy.
* History of invasive surgery for glaucoma (including laser therapy).
* Anterior segment or intraocular surgery (other than glaucoma) within 90 days prior to start of washout phase.
* History of severe eye injury.
* History of allergy to agents that were to be used during the study (e.g., benzalkonium chloride, instillation anesthetics, fluorescein, latanoprost eye drops).
* Intended use of prohibited concomitant medications or therapies during the study.
* Required use of contact lenses from 1 week before treatment phase initiation and during the study.
* Pseudophakic eye, aphakic eye.
* Current participation in another clinical study, or participation and treatment with study medication within 90 days before the start of the washout phase.
* Females who are pregnant, nursing, or potentially pregnant (e.g., positive pregnancy test), planning a pregnancy during the study, or unable to use appropriate contraception during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Intraocular Pressure (IOP) at Week 4 | Week 4
  Change from Baseline in Mean Diurnal IOP at Week 4

SECONDARY OUTCOMES:
Percent Change in Intraocular Pressure (IOP) | Week 4
  Percent Change from Baseline in Mean Diurnal Intraocular Pressure (IOP) at Week 4
Change and Percent Change in Intraocular Pressure (IOP) | Post baseline Visits except Week 4
  Change and Percent Change from Baseline in Mean Diurnal IOP at each post baseline visit except week 4.
Change and Percent Change from baseline in Intraocular Pressure (IOP) | Assessment time point at each post baseline visit.
  Change and Percent Change from baseline in IOP at each IOP assessment time point at each post baseline visit.
Percentage of Responders | Each Post Baseline Visit.
  Percentage of Responders (percent reduction from baseline in Mean Diurnal IOP: ≥20%, ≥25%, ≥30%) at each post baseline visit.

CONTACTS AND LOCATIONS:
Locations (25):
- China (25):
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing
  - Beijing Hospital, Beijing
  - Beijing Tongren Hospital, Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Zhongshan Ophthalmic Center, Guangzhou
  - Affiliated Hospital of Guizhou Medical University, Guiyang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Jinan Second People's Hospital (Jinan eye hospital), Jinan
  - The Second Hospital & Clinical Medicial Lanzhou University, Lanzhou
  - Luoyang third people's hospital, Luoyang
  - Qingdao Eye Hospital of Shandong First Medical University, Qingdao
  - Shanghai Eye Disease Prevention And Treatment Center/Shanghai Eye Hospital, Shanghai
  - Joint Shantou International Eye Center of Shantou University and the Chinese University of Hong Kong, Shantou
  - Shanxi eye hospital, Shanxi
  - Aier Eye Hospital (Liaoning), Shenyang
  - The 4th People's Hospital of Shenyang, Shenyang
  - Shenzhen Eye Hospital, Shenzhen
  - Tianjin Eye Hospital, Tianjin
  - Weifang Eye Hospital, Weifang
  - Wuhan Aier Eye Hospital, Wuhan
  - Wuhan Puren Hospital, Wuhan
  - Zhongnan Hospital Affiliated to Wuhan University, Wuhan
  - Wuxi Second People's Hospital, Wuxi
  - Xiamen Eye Centre of Xiamen University Co., Ltd., Xiamen

IPD SHARING:
Plan to Share IPD: No